CLINICAL TRIAL: NCT00533130
Title: Phase 2/3 Eficacy Study of the AO Pediatric Classification in Treatment and Prognosis of Long Bones Fractures
Brief Title: Evaluation of the AO Pediatric Classification for Long Bones Fractures Like a Guide for Treatment and Prognosis
Acronym: AO-PC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Cruz Roja Mexicana (Other)
Other Study IDs: CRM-2008-TYO
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Fractures; Children
Keywords: AO; Pediatric; Classification; Long Bones; fractures; bones
MeSH Terms: conditions — Fractures, Bone | interventions — Observation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Pediatric patients under 16 years old with long bones fractures
  Interventions: Procedure: clinical evaluation; Procedure: observational study

INTERVENTIONS:
Procedure: clinical evaluation — analyze the x ray from each patient and evaluate the treatment y development of bone healing.
  Other Names: AO classification
Procedure: observational study — evaluate the walk patron, bone healing and range of motion at 1,3,6,12 months
  Other Names: AO clasification

SUMMARY:
1. Is the AO Pediatric classification for long bones fractures reproductible?
2. Is the AO Pediatric Classification for long bones fractures a treatment guide?
3. The AO pediatric Classification for long bones fractures could be a prognosis factor?

DETAILED DESCRIPTION:
PROPOUSE:

1. To determinate the efectivity of the AO pediatric classification for long bones fractures.
2. To evaluate the functionality of the AO pediatric classification for long bones fractures.
3. To analyze if the AO pediatric classification for long bones fractures is a prognosis factor

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Less than 16 years old.
* Open physis.
* Long bone fractures.
* X ray AP & lateral comparatives.
* Informed consent for parents or tutor.
* Don´t let the treatment during the time of study.

Exclusion Criteria:

* Pathologic fractures.
* Fractures not included en the AO pediatric classification for long bones.
* Diseases that modifying the bone healing: Diabetes mellitus, osteogenesis imperfect, etc.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge D Tejada-Hoyos, M.D., Principal Investigator — orthopaedic resident
Locations (1):
- Hospital Cruz Roja Mexicana, Delegacion Distrito Federal, Mexico City, Federal District, Mexico